CLINICAL TRIAL: NCT01889043
Title: Monitoring of Non-invasive Ventilation During Sleep in ALS
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Dries Testelmans, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S53536
Record Dates: First submitted 2013-05-07; First posted 2013-06-28 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Noninvasive Ventilation; Polysomnography
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-invasive ventilation (NIV) has already shown to improve survival and quality of life in patients with amyotrophic lateral sclerosis (ALS). Quality of sleep seems already to be impaired in patients with preserved diaphragmatic dysfunction. Until now, only few research has been performed on the quality of sleep in patients with ALS when using NIV, and these data are mainly based on patient reported outcomes.Further on, only very little research has been done on patient-ventilator interaction.

Our study would like to perform research on quality of sleep before and after NIV use by using full polysomnography with incorporation of transcutaneous carbon dioxide measurement and built-in ventilator software.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ALS (according to El Escorial criteria) who are planned to start to use NIV, objectivated by a decreased inspiratory muscle force with a restrictive pulmonary function and

  1. symptoms of nocturnal alveolar hypoventilation or
  2. increased daytime arterial carbon dioxide partial pressure (PCO2)(> 45 mmHg) or
  3. a ≥ 10 mmHg increase in transcutaneous PCO2 during sleep in comparison to a normal awake supine value

Exclusion Criteria:

* Patients < 18 years
* Patients not willing to start NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Amyotrophic lateral sclerosis patients, which are followed at the Neuromuscular Reference Centre UZ Leuven, in need for NIV treatment
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in transcutaneous carbon dioxide and respiratory events | At day 2, 3 and 4 and at 1, 3, 6, 9 and 12 months
  Search for an optimal titration protocol. Aim is to reduce transcutaneous carbon dioxide (CO2) below 55 mmHg and to reduce central and obstructive respiratory events to a minimum. This will be assessed by performance of a nocturnal measurement of transcutaneous CO2 and full polysomnography at eacht time point.
Change in patient-ventilator asynchronies | Day 4 and at 1,3,6,9 and 12 months
  The following asynchronies will be evaluated: auto-triggering, double triggering, ineffective effort, prolonged insufflation. The impact of leaks will also be evaluated.Data will be reported as events/hour of sleep. This will be assessed by full polysomnography at each time point.

SECONDARY OUTCOMES:
Impact of NIV on sympatho-vagal balance | Day 1 and at 1,3,6,9 and 12 months
changes in quality of life by patient reported outcomes | Day 1 and at 1,3,6,9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dries Testelmans, MD,PhD, Principal Investigator — UZ Leuven; Bertien Buyse, MD, PhD, Study Director — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium